CLINICAL TRIAL: NCT00644384
Title: Chemoprevention Trial of Acitretin Versus Placebo in Patients at High Risk for Basal Cell Carcinoma or Squamous Cell Carcinoma
Brief Title: Acitretin in Preventing Skin Cancer in Patients at High Risk for Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mark R Pittelkow, M.D., Mayo Clinic
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000582327; P30CA015083 (NIH); MC02C8 (Other: Mayo Clinic Cancer Center); 1153-98 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-22; First posted 2008-03-26 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Acitretin; Gene Expression Profiling; Blotting, Northern; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: acitretin
Genetic: gene expression analysis
Genetic: northern blotting
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of acitretin may stop cancer from growing in patients at high risk for basal cell carcinoma or squamous cell carcinoma of the skin.

PURPOSE: This randomized trial is studying how well acitretin works in preventing skin cancer in patients at high risk for skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the chemopreventive efficacy of acitretin, a synthetic retinoid, in patients at high risk for basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin.
* Evaluate human papillomavirus (HPV) as a possible etiologic cofactor in the development of cutaneous epidermal dysplasia/carcinoma from skin tissues of patients at high risk for BCC or SCC of the skin.
* Determine the effect of acitretin on a series of potential surrogate endpoint biomarkers (SEBs), including specific retinoid receptors; the Fos/Jun family of proto-oncogenes and products; the Fos/Jun family of transcription factor complexes known as activating protein 1 (AP-1); and HPV DNA in normal (sun-protected), sun-exposed dysplastic and carcinoma (SCC/BCC) skin specimens.
* Correlate standard clinical and histopathological dermatologic evaluation with modulation of SEBs.

OUTLINE: This is a multicenter study. Patients are stratified according to age (18-49 years vs 50-59 years vs 60-69 years vs ≥ 70 years), number of skin cancers within the past 5 years (2-5 vs 6-10 vs 11-20 vs 21-30 vs > 30), most recent skin cancer occurrence (< 12 months ago vs ≥ 12 months ago), patient-reported sunburn susceptibility by Fitzpatrick skin type (1 vs 2 vs 3 vs 4 vs 5 vs 6), and assessment of visible skin damage (minimal vs moderate vs extensive). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral acitretin 5 days a week for 2 years in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo 5 days a week for 2 years in the absence of unacceptable toxicity.

Tissue samples of normal skin, excised squamous cell or basal cell carcinoma, or excised actinic keratoses are obtained at baseline and periodically during study. Tissue samples are analyzed for surrogate endpoint biomarkers, including RARγ, RXRα, Fos/Jun family of proto-oncogenes and products, AP-1 DNA binding activity, and presence, identification, and quantification of HPV DNA. mRNA and protein expression levels of RARγ, RXRα, and Fos/Jun family members are analyzed by northern blotting and/or quantitative polymerase chain reaction (PCR) methods. HPV is analyzed by PCR.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin, defined as a prior history of ≥ 3 nonmelanoma skin lesions

  * All visible BCC or SCC must have been resected prior to study entry

PATIENT CHARACTERISTICS:

* Life expectancy > 5 years
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* SGOT ≤ 2 times ULN
* Creatinine ≤ 1.5 times ULN
* Cholesterol < 250 mg/dL
* Triglycerides < 2.5 times ULN
* Not pregnant
* No history of significant, uncontrolled hyperlipidemia
* No history of oral retinoid intolerance
* No history of other significant medical condition that, in the opinion of the physician, would contraindicate retinoid use

PRIOR CONCURRENT THERAPY:

* More than 1 year since prior retinoid therapy
* At least 4 weeks since prior and no other concurrent use of oral vitamin A supplements, topical retinoids, or other potentially irritating skin preparations

  * Concurrent multivitamin supplements allowed
* No prior organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2003-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Rate of new non-melanoma skin cancer development

SECONDARY OUTCOMES:
Time to new non-melanoma skin cancer development
Gene expression (RAR/RXR, Fos/Jun, and AP-1)
HPV DNA detection, sequencing, and quantification

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Pittelkow, MD, Principal Investigator — Mayo Clinic